CLINICAL TRIAL: NCT00881998
Title: Prospective, Randomized Study of Two Surgical Approaches for Total Hip Arthroplasty
Brief Title: Study of Two Surgical Approaches for Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Rothman Institute Orthopaedics
Allocation: Randomized | Purpose: Treatment
Other Study IDs: RIUWHOZ-09-02
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Last update posted 2009-04-16 (Estimated); Status verified 2009-04

CONDITIONS: Total Hip Arthroplasty
Keywords: Evaluate early functional outcomes of two anterior approaches to total hip arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Minimally invasive total hip arthroplasty
  Interventions: Procedure: Minimally Invasive Total Hip Arthroplasty
- 2 (Active Comparator)
  Interventions: Procedure: Conventional Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Minimally Invasive Total Hip Arthroplasty
  Arms: 1
Procedure: Conventional Total Hip Arthroplasty
  Arms: 2

SUMMARY:
A prospective, comparative, randomized single surgeon study comparing minimally invasive total hip arthroplasty (MIS) via anterior approach to conventional total hip arthroplasty via anterolateral transgluteal approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with osteoarthritis of the hip and have decided to undergo total hip arthroplasty
* Patients willing to sign the consent form

Exclusion Criteria:

* Patient is unwilling to sign the consent form
* Patient is involved in another study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Hozack, MD, Principal Investigator — Rothman Institute Orthopaedics
Locations (1):
- Rothman Institute Orthorpaedics, Philadelphia, Pennsylvania, United States